CLINICAL TRIAL: NCT00993369
Title: Heart Rate Variability in Children Conceived Via Assisted Reproductive Technologies
Acronym: HRV ART
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 00018811
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Neuro Developmental Delay
Keywords: Prediction of neuro developmental delay

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy newborns conceived naturally
  Interventions: Other: Holter monitor
- Healthy newborns conceived with IVF
  Interventions: Other: Holter monitor

INTERVENTIONS:
Other: Holter monitor — Record heart rate for 2 to 6 hours on day of life 1 or 2.

SUMMARY:
This is a proof of principle study that investigates heart rate variability differences in fetal and neonatal life in a longitudinal study design and compares two subject groups, offspring conceived using in-vitro fertilization and conceived naturally.

DETAILED DESCRIPTION:
This is a proof of principle study that investigates heart rate variability differences in fetal and neonatal life in a longitudinal study design and compares two subject groups, offspring conceived using in-vitro fertilization and conceived naturally.

ELIGIBILITY:
Inclusion Criteria:

* Fetus or newborn
* Delivery at University of Utah Medical Center, Latter Day Saints Hospital or Intermountain Medical Center

Exclusion Criteria:

* Twins
* Genetic anomaly
* Congenital malformation
* Need for special care

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fetus and newborns.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability in Children Conceived Via Assisted Reproductive Technologies | 2 to 6 hours
  Holter monitor/2 aims

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Medical Center, Salt LakeCity, Utah, United States